CLINICAL TRIAL: NCT04906512
Title: A Randomized Perspective, Open and Parallel Controlled Study Comparing 3M Tegaderm CHG I.V. Securement Dressing With 3M Tegaderm Transparent Dressing for Evaluation of Antimicrobial Efficacy on DVC Insertion Site in Adult in Critical Care
Brief Title: Comparing CHG I.V. Securement Dressing With Transparent Dressing for Evaluation of Antimicrobial Efficacy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The decision to terminate this clinical study was made as a cost control measure.
Sponsor: Solventum US LLC (Industry)
Collaborators: 3M (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EM-05-014894
Record Dates: First submitted 2021-01-14; First posted 2021-05-28 (Actual); Results first posted 2023-10-06 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Central Venous Catheter Exit Site Infection; Catheter-Related Infections
MeSH Terms: conditions — Catheter-Related Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- 3M™ Tegaderm™ CHG I.V. Securement Dressing (Experimental): The primary purpose of 3M™ Tegaderm™ CHG I.V. Securement Dressing is to secure devices to skin; and secondly, the dressing contains an antimicrobial ingredient that inhibits microbial regeneration. This product is used to cover and protect the catheter sites on the body surface and to secure devices to skin and is available in a variety of models and sizes.
  Interventions: Device: 3M™ Tegaderm™ CHG I.V. Securement Dressing
- 3M™ Tegaderm™ Transparent Film Dressing 1626W (Active Comparator): Transparent dressing, i.e. CHG-free transparent dressing, can be used to cover and protect catheter sites on the body surface and to secure devices to skin, without any antibacterial ingredients, and are the currently most commonly used transparent dressings in DVC care in China.
  Interventions: Device: 3M™ Tegaderm™ Transparent Film Dressing 1626W

INTERVENTIONS:
Device: 3M™ Tegaderm™ CHG I.V. Securement Dressing — Subjects eligible for enrollment will be randomly assigned to either the Tegaderm CHG dressing group or the transparent dressing group, and patients in both groups will be given catheterization according to the hospital's standards and nursed according to the catheter maintenance procedure. The investigator would monitor the subjects during dressing changes, observing the subjects' general conditions, skin condition at the DVC site and the dressing condition, and change a dressing or take relevant measures (if applicable), until the end of the trial, i.e. CVC removal or patient transfer out of the ICU.
  Arms: 3M™ Tegaderm™ CHG I.V. Securement Dressing
Device: 3M™ Tegaderm™ Transparent Film Dressing 1626W — Subjects eligible for enrollment will be randomly assigned to either the Tegaderm CHG dressing group or the transparent dressing group, and patients in both groups will be given catheterization according to the hospital's standards and nursed according to the catheter maintenance procedure. The investigator would monitor the subjects during dressing changes, observing the subjects' general conditions, skin condition at the DVC site and the dressing condition, and change a dressing or take relevant measures (if applicable), until the end of the trial, i.e. CVC removal or patient transfer out of the ICU.
  Arms: 3M™ Tegaderm™ Transparent Film Dressing 1626W

SUMMARY:
This is a single-center, prospective, randomized controlled clinical trial designed to compare the antimicrobial efficacy of Tegaderm CHG I.V. Securement Dressing and transparent dressings for deep vein catheterization in adult ICU patients.

DETAILED DESCRIPTION:
This clinical trial is designed as a prospective, randomized, open-label, parallel-group controlled trial.

Investigational product: 3M™ Tegaderm™ CHG I.V. Securement Dressing Control product: 3MTM TegadermTM Transparent Film Dressing 1626W

Considering the easy-to-distinguish appearances of both products used, this trial will adopt an open-label design. The primary endpoint is the rate of CVC tip colonization (positive catheters after culture/total catheters).

Subjects eligible for enrollment will be randomly assigned to either the Tegaderm CHG dressing group or the transparent dressing group, and patients in both groups will be given catheterization according to the hospital's standards and nursed according to the catheter maintenance procedure. The investigator would monitor the subjects during dressing changes, observing the subjects' general conditions, skin condition at the DVC site and the dressing condition, and change a dressing or take relevant measures (if applicable), until the end of the trial, i.e. CVC removal or patient transfer out of the ICU.

440 subjects who meet the inclusion/exclusion criteria will be enrolled. Subjects will be adult voluntary clinical subjects, of either sex, at least 18 years of age, who are ICU patients undergoing deep venous catheterization (DVC), in which a CVC catheter must be used while other types of catheters such as hemodialysis, PICCO, and floating catheters may be used concurrently.

ELIGIBILITY:
Inclusion Criteria:

Subjects may be included that meet the following criteria:

1. Subjects should be at least 18 years old or older at the time of providing consent;
2. Subjects would be available to attend all visits required in the trial, be inpatients in the Department of Critical Care Medicine and have an expected length of stay in the ICU of no less than 3 days;
3. The subject or his/her legally authorized representative should be competent to sign the informed consent form;
4. The patient must have a central venous catheter (CVC) used on him/her, which may or may not be used in combination with other types of DVCs;
5. The patient's catheter insertion site is free of deformities, phlebitis, infiltrations, dermatitis, eczema, rashes, breaks, burns, tattoos or other skin conditions that may affect the integrity of the skin at the insertion site;
6. The patient would comply with the DVC treatment process and the nursing process prescribed in this protocol.

Exclusion Criteria:

Subjects may not be included that meet any of the following criteria:

1. The subject is unwilling/unable to attend study visits (unlike IC);
2. There is sunburn, skin infection or scar, mole or other blemishes on the subject's catheterization site that would affect the scoring or measurement of the site;
3. The patient is assessed by the investigator as being at high risk of CLABSI, or known to be CLABSI, based on the environment, duration, and site conditions of catheterization;
4. The patient is documented or known to have allergies (sensitivities) to adhesive products, or other products involved in the trial, e.g. transparent dressings, CHG and alcohol;
5. The patient is being or has been subjected to other antibiotic, catheter or skin-related clinical trials;
6. The patient needs topical application of creams containing antimicrobial ingredients or other antimicrobial fluids beneath the Tegaderm CHG dressing or transparent dressing for skin disinfection, in addition to the requirements of this protocol;
7. The patient is assessed by the investigator as being at high risk of blood stream infection, or known to be sepsis, caused by blood stream infection;
8. The patient has dermatitis, burns, lesions, breaks, eczema, tattoos or other conditions at the catheter insertion site that would interfere with observation in the trial;
9. Women who are pregnant or breast feeding;
10. Patients who are not eligible for the study at the discretion of other investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2021-05-14 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hongping Qu, Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: After 123 subjects were enrolled and completed all the visits, the study was terminated.
Period: Overall Study
Arm/Group | 3M™ Tegaderm™ Transparent Film Dressing 1626W | 3M™ Tegaderm™ CHG I.V. Securement Dressing
Started | 62 | 61
Completed | 39 | 42
Not Completed | 23 | 19

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 3M™ Tegaderm™ CHG I.V. Securement Dressing | 3M™ Tegaderm™ Transparent Film Dressing 1626W | Total
Number analyzed (Participants) | 61 | 62 | 123
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.5 (16.84) | 66.4 (12.88) | 65.4 (14.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 18 | 36
  Male | 43 | 44 | 87
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 61 | 62 | 123
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 61 | 62 | 123

OUTCOME MEASURES:

1. Primary Outcome: Rate of CVC Tip Colonization (Positive Catheters After Culture/Total Catheters)
Description: Rate of CVC tip colonization (positive catheters after culture/total catheters)
Time Frame: 3-14 days
Population: This endpoint was not collected for all subjects randomized. Also, the study had major protocol deviations that made the available data unreliable.
Arm/Group | 3M™ Tegaderm™ Transparent Film Dressing 1626W | 3M™ Tegaderm™ CHG I.V. Securement Dressing
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 3-14 days
Arm/Group | 3M™ Tegaderm™ Transparent Film Dressing 1626W | 3M™ Tegaderm™ CHG I.V. Securement Dressing
All-Cause Mortality (participants affected / at risk) | 2/62 | 0/61
Serious Adverse Events (participants affected / at risk) | 2/62 | 0/61
Other Adverse Events (participants affected / at risk) | 44/62 | 46/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 3M™ Tegaderm™ Transparent Film Dressing 1626W (N=62) | 3M™ Tegaderm™ CHG I.V. Securement Dressing (N=61)
Circulatory collapse (Vascular disorders) | 1 (1) | 0 (0)
Intraventricular hemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 3M™ Tegaderm™ Transparent Film Dressing 1626W (N=62) | 3M™ Tegaderm™ CHG I.V. Securement Dressing (N=61)
Heart rate increased (Investigations) | 6 | 5
Pyrexia (General disorders) | 14 | 15
Hypoproteinaemia (Metabolism and nutrition disorders) | 10 | 5
Hypertension (Vascular disorders) | 5 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 3 | 2
Amylase increased (Investigations) | 3 | 0
Hypotension (Vascular disorders) | 2 | 3
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 3
Haematuria (Renal and urinary disorders) | 0 | 3
Delirium (Psychiatric disorders) | 0 | 3
Blood bilirubin increased (Investigations) | 2 | 2
White blood cell count increased (Investigations) | 2 | 1
Aspartate aminotransferase increased (Investigations) | 2 | 1
Blood pressure increased (Investigations) | 2 | 1
Oxygen saturation decreased (Investigations) | 1 | 2
Blood creatinine increased (Investigations) | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 2
Vomiting (Gastrointestinal disorders) | 0 | 2
Atrial fibrillation (Cardiac disorders) | 1 | 2
Incision site haemorrhage (Injury, poisoning and procedural complications) | 0 | 2
Incision site discharge (Injury, poisoning and procedural complications) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-04-05): https://cdn.clinicaltrials.gov/large-docs/12/NCT04906512/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-25): https://cdn.clinicaltrials.gov/large-docs/12/NCT04906512/SAP_001.pdf